CLINICAL TRIAL: NCT06558604
Title: A Phase II, Multicenter, Open-label Study Evaluating Glofitamab in Combination With Venetoclax Plus Zanubrutinib or Venetoclax Alone in Subjects With Untreated or Relapsed/Refractory High-risk Mantle-cell Lymphoma
Brief Title: Phase II Study of Glofitamab With Venetoclax +/- Zanubrutinib in High-risk Mantle-cell Lymphoma
Acronym: GLOASIS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: BeiGene (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLOASIS
Record Dates: First submitted 2024-07-24; First posted 2024-08-16 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Lymphoma, Mantle-Cell
Keywords: POD24; BTKI failure; High risk; 18 to 79 years
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — obinutuzumab; glofitamab; zanubrutinib

STUDY DESIGN:
Intervention Model Description: 3 cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A - POD24 (Experimental): * Obinutuzumab IV infusion 2000 mg flat dose at C1D1 or Splited in 2 doses of 1000 mg at C1D1 and C1D2
  * Glofitamab IV infusion 2.5 mg C1D8 10 mg C1D15 30 mg C2D1 and C3D1 (infusion during min 4 hours ) 30 mg Each D1 for C4 to C6 (Infusion during min 2 hours ) 30 mg Each D1 for C7 to C12 (Infusion during min 90 min)
  * Zanubrutinib PO 320 mg total daily dose (QD) From C1D2 continuously until end C35
  * Venetoclax PO 20 mg/d C2D3 to C2D7 50 mg/d C2D8 to C2D14 100 mg/d C2D15 to C2D21 200 mg/d C3D1 to C3D7 400 mg/d From C3D8 continuously until end C35
  Interventions: Drug: Obinutuzumab; Drug: Glofitamab; Drug: Venetoclax Oral Product
- Cohort B - BTKI failure (Experimental): * Obinutuzumab IV infusion 2000 mg flat dose at C1D1 or Splited in 2 doses of 1000 mg at C1D1 and C1D2
  * Glofitamab IV infusion 2.5 mg C1D8 10 mg C1D15 30 mg C2D1 and C3D1 (infusion during min 4 hours ) 30 mg Each D1 for C4 to C6 (Infusion during min 2 hours ) 30 mg Each D1 for C7 to C12 (Infusion during min 90 min)
  * Venetoclax PO 20 mg/d C2D3 to C2D7 50 mg/d C2D8 to C2D14 100 mg/d C2D15 to C2D21 200 mg/d C3D1 to C3D7 400 mg/d From C3D8 continuously until end C35
  Interventions: Drug: Obinutuzumab; Drug: Glofitamab; Drug: Venetoclax Oral Product
- Cohort C - first Line (Experimental): * Obinutuzumab IV infusion 2000 mg flat dose at C1D1 or Splited in 2 doses of 1000 mg at C1D1 and C1D2
  * Glofitamab IV infusion 2.5 mg C1D8 10 mg C1D15 30 mg C2D1 and C3D1 (infusion during min 4 hours ) 30 mg Each D1 for C4 to C6 (Infusion during min 2 hours ) 30 mg Each D1 for C7 to C12 (Infusion during min 90 min)
  * Zanubrutinib PO 320 mg total daily dose (QD) From C1D2 continuously until end C35
  * Venetoclax PO 20 mg/d C2D3 to C2D7 50 mg/d C2D8 to C2D14 100 mg/d C2D15 to C2D21 200 mg/d C3D1 to C3D7 400 mg/d From C3D8 continuously until end C35
  Interventions: Drug: Obinutuzumab; Drug: Glofitamab; Drug: Venetoclax Oral Product; Drug: Zanubrutinib Oral Capsule

INTERVENTIONS:
Drug: Obinutuzumab — 1000 mg/40mL
  Other Names: Gazyvaro
Drug: Glofitamab — 10mg/mL
  Other Names: Columvi 10 mg
Drug: Venetoclax Oral Product — 10mg, 50mg and 100mg tablets
  Other Names: Venclyxto
Drug: Zanubrutinib Oral Capsule — 80mg capsules
  Other Names: Zanubrutinib (BGB-3111)
  Arms: Cohort C - first Line

SUMMARY:
This open-label, multicenter, three cohorts, phase II study is designed to assess a combination of Zanubrutinib/Venetoclax/Glofitamab or Venetoclax/Glofitamab in high-risk subjects with either first line or R/R Mantle Cell Lymphoma (MCL).

Three independent cohorts will be run:

* Cohort A will include subjects with a primary refractory or progressive disease within 24 months from initiation of first line treatment (POD 24).
* Cohort B will be open for subjects with R/R MCL and refractory or progressive to a BTK inhibitor given previously (>24 months if first line).
* Cohort C will only enrol newly diagnosed and untreated MCL subjects with very high-risk features.

DETAILED DESCRIPTION:
Cohort A : 40 subjects will be included and treated Cohort B : 36 subjects will be included and treated Cohort C : 24 subjects will be included and treated

Subjects in cohorts A and C will receive during induction phase 12 cycles of Zanubrutinib/Venetoclax/Glofitamab and during maintenance phase 23 cycles of Zanubrutinib/Venetoclax

Subjects in cohort B will receive during induction phase 12 cycles of Venetoclax/Glofitamab and during maintenance phase 23 cycles of Venetoclax

ELIGIBILITY:
Inclusion Criteria:

In cohort A, subject must meet the following inclusion criteria:

1. Subject must be primary refractory or in progression within 24 months from initiation of first line treatment (POD24 defined as time between D1C1 of the first treatment line and ICF signature)) (including an anti-CD20 combined with chemotherapy). Subject previously exposed to BTK inhibitor at first line is eligible. Subject in failure of CAR-T cell first line is eligible.
2. Primary refractory subjects (ie with a progressive disease) to the BTKi and Venetoclax combination will not be eligible.

   In cohort B, subject must meet the following inclusion criterion:
3. Subject must be R/R MCL and refractory or progressive to a BTK inhibitor given in a previous line of treatment (the number of treatment lines is not limited). If first progression, time from diagnosis (defined as D1C1 of the first treatment line) to inclusion (defined as the date of ICF signature) must be superior to 24 months.
4. Subject previously exposed to Bcl-2 therapy and/or relapsing post CAR-T cell therapy is eligible, except if they presented a progressive disease under BTKi and Venetoclax combination.

   In cohort C, subject must meet the following inclusion criteria:
5. Subject not previously treated for mantle cell lymphoma.
6. Subject at high risk of relapse presenting at least two of the following risk factors:

   1. TP53 mutation, del17p, or p53 expression (IHC) > 50%,
   2. blastoïd variant,
   3. complex karyotype,
   4. c-myc rearrangement (FISH),
   5. Ki67≥30%,
   6. high MIPI score, (or MIPI simplified)
   7. high MIPI-combined score ((ie high MIPI score + Ki67≥30%): this criterion alone is sufficient.

   Subject must meet all of the following additional criteria to be enrolled in the study for cohort A, B and C:
7. Subject is ≥ 18 years and < 80 years of age at the time of signing the informed consent form (ICF).
8. Subject understood and voluntarily signed and dated an informed consent prior to any study-specific assessments/procedures being conducted.
9. Subject with histologically proven mantle cell lymphoma (latest WHO classification). The diagnosis has to be confirmed by phenotypic expression of CD5, CD20 and cyclin D1 or the t(11;14) translocation. Diagnostic tissue should be available for central pathology review and ancillary molecular studies.
10. Bi-dimensionally measurable disease defined by at least one single node or tumor lesion ≥ 1.5 cm assessed by CT scan, or one bi-dimensionally measurable (≥1 cm) extranodal lesion, as measured on CT scan, and/or clinical examination.
11. Stage II-IV disease,
12. ECOG performance status of 0, 1, 2.
13. Life expectancy of more than 3 months.
14. Adequate renal function as demonstrated by a creatinine clearance > 30 mL/min; calculated by the Cockcroft Gault formula or MDRD formula.
15. Adequate hepatic function per local laboratory reference range as follow (unless if due to lymphoma involvement):

    1. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5x upper limit of normal (ULN)
    2. Bilirubin < 1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin. in which case total bilirubin should be < 3 x ULN).
16. Women of childbearing potential (WOCBP) (refer to section 14.7 for more details) must have negative results for highly effective urine/serum pregnancy test 10-14 days prior to Day 1 of Cycle 1 and within 24 hours prior to day 1 Cycle 1 prior to initiating study treatment and agree to abstain from becoming pregnant or breastfeeding during study participation and until at least 18 months after C1 with Obinutuzumab, or 3 months after the final dose of tocilizumab (if applicable), or 2 months after the final dose of Glofitamab, or or 1 month after the final dose of Zanubrutinib (if applicable), or 30 days after the final dose of Venetoclax, whichever is longer. WOCBP agree to remain abstinent (from heterosexual intercourse) or use two methods of contraception, and to refrain from donating eggs, during the treatment period and for at least 18 months after the final dose of Obinutuzumab, 3 months after the final dose of tocilizumab (if applicable), 2 months after the final dose of Glofitamab, 1 month after the final dose of Zanubrutinib (if applicable), and 30 days after the final dose of Venetoclax (refer to section 14.6).
17. Men of reproductive potential (refer to section 14.6 for more details) agree to remain abstinent (from heterosexual intercourse) or use effective methods of birth control with a non-pregnant female partner of childbearing potential or a pregnant female partner and to refrain from donating sperm, during the treatment period and for at least 3 months after the final dose of Obinutuzumab, 2 months after the final dose of Glofitamab, 2 months after the final dose tocilizumab (if applicable), 30 days after the final dose of Venetoclax, 1 week after the final dose of Zanubrutinib (if applicable).
18. Adequate bone marrow function as defined by:

    1. Absolute neutrophil count (ANC) ≥ 1000/mm3, except for subjects with bone marrow involvement in which ANC must be ≥ 500/mm3.
    2. Platelet ≥ 75,000/mm3, except for subjects with bone marrow involvement in which the platelet count must be ≥ 50,000/mm3 .
19. Subject covered by any social security system (France).
20. Subject who understands and speaks one of the country official languages unless local regulation authorizes independent translators.
21. Subject with a SARS-COV2 vaccination status in line with local National guidelines/recommendations (COSV, ANRS MIE).
22. Subject must be willing and able to comply with protocol-mandated hospitalization upon administration of the first two doses of Glofitamab. Subject must also be willing to comply with all study-related procedures.
23. Adverse events from prior anti-cancer therapy must have resolved to Grade ≤ 1 (hematological toxicities excepted)

    -

Exclusion Criteria:

Subject who meets any of the following criteria will be excluded from enrollment in the study study for cohort A, B and C:

1. Proven or previously known CD20 negative status on FFPE IHC at time of MCL relapse or diagnosis.
2. For subjects in Cohort A and B: previously refractory to treatment by BTK inhibitor and Bcl-2 therapy combination.
3. Any prior therapy with a bispecific antibody targeting CD3 and CD20.
4. Current or past history of central nervous system or meningeal involvement by lymphoma.
5. Use of any standard or experimental anti-cancer drug therapy including biological agents (e.g. monoclonal antibodies) within 30 days of the start (Day 1) of study treatment, except for BTKi for subjects included in cohort B, that can be pursued until C1D1. and except for topical treatment or hormone treatment if criterion 33 is respected. Corticosteroid treatment ≤ 1 mg/kg/day prednisone or equivalent is allowed within 2 weeks prior to Obinutuzumab infusion.
6. LVEF < 50% as determined by echocardiography or isotopic method.
7. Clinically significant cardiovascular disease such as uncontrolled, unstable or symptomatic arrhythmias, unstable angina, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class III (moderate) or Class IV(severe) cardiac disease as defined by the New York Heart Association Functional Classification or Objective Assessment Class C or D cardiac disease. Heart rate-corrected QT interval > 480 milliseconds based on Fridericia's formula.; History of Mobitz II second-degree or third-degree heart block without a permanent pacemaker in place; Uncontrolled hypertension as indicated by a minimum of 2 consecutive blood pressure measurements, at screening, showing systolic blood pressure > 170 mmHg and diastolic blood pressure > 105 mmHg and/or uncontrolled hypertension with systolic blood pressure>140mmHg despite a well conduct hypertensive treatment for at least 6 months
8. Hemoglobin level < 8g/dL; Absolute Neutrophil count <1 G/L (<0,5G/L if related to lymphoma); Platelets < 75 G/L (< 50 G/L if related to lymphoma),
9. Major surgery within 28 days before screening.
10. Require the use of anticoagulation by warfarin or equivalent vitamin K antagonists (e.g., phenprocoumone)
11. Requires treatment with a moderate or a strong CYP3A inhibitor or inducer..
12. Vaccinated with live, attenuated vaccines within 4 weeks of enrollment (except COVID vaccine) or anticipation that such a live attenuated vaccine will be required during the study.
13. Known hypersensitivity to active substances or to any of the excipients. Or Contraindication to any study treatments.
14. Known allergy to all xanthine oxidase inhibitors or rasburicase.
15. Previously documented G6DP deficiency.
16. Severe prior reactions to anti CD20 monoclonal antibodies or prior significant toxicity (other than thrombocytopenia) with Bcl-2 inhibitor.
17. Prior treatment with systemic immunosuppressive medications (including, but not limited to, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents), within 2 weeks or five half-lives (whichever is shorter) prior to first dose of study treatment.
18. Unable to swallow capsules or disease significantly affecting gastrointestinal function such as malabsorption syndrome, resection of the stomach or small bowel, bariatric surgery procedures, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
19. History of severe bleeding disorder such as hemophilia A, hemophilia B, von Willebrand disease, or history of spontaneous bleeding requiring blood transfusion or other medical intervention.
20. Current or history of CNS disease, such as stroke, epilepsy, CNS vasculitis, neurodegenerative disease: or intracranial hemorrhage: Subjects with a history of stroke or intracranial hemorrhage who have not experienced a stroke or transient ischemic attack or intracranial hemorrhage within the past 2 years and have no residual neurologic deficits, as judged by the investigator, are allowed.
21. Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment or any major episode of infection (as evaluated by the investigator) within 4 weeks prior to the first study treatment.
22. Known Human Immunodeficiency Virus (HIV), for subjects with unknown HIV status, HIV testing will be performed at screening if required by local regulations.
23. Positive test results for hepatitis C virus (HCV) antibody: Subjects who are positive for HCV antibody are eligible only if PCR is negative for HCV RNA.
24. Positive test results for hepatitis B virus (HBV) infection (defined as positive HbsAg serology) Subjects with occult or prior HBV infection (defined as negative HbsAg and positive HbcAb) may be included if HBV DNA is undetectable, provided that they are willing to undergo DNA testing on Day 1 of every cycle and every three months for at least 12 months after the last cycle of study treatment and appropriate antiviral therapy.
25. Positive SARS-CoV-2 test within 7 days prior to enrollment. Rapid antigen test result is also acceptable.
26. Documented SARS-CoV-2 infection within 6 months of first study treatment (Cycle 1 Day 1): Subjects may be eligible if they have no persistent respiratory symptoms, no evidence of lung infiltrates on chest CT, and have a negative PCR during the first 30 days prior to first study treatment (Cycle 1 Day 1)
27. Suspected or latent tuberculosis (confirmed by positive interferon-γ release assay)
28. Known or suspected chronic active Epstein-Barr viral infection.
29. Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator opinion, could compromise the subject's safety, interfere with the absorption or metabolism of study treatments, or put the study outcomes at undue risk.
30. Prior allogenic SCT is allowed if no active GVHD and no active immune-suppressive treatment (to be discussed with the medical monitor).
31. Active autoimmune disease requiring treatment:

    1. Subjects with a history of autoimmune-related hypothyroidism on a stable dose of thyroid-replacement hormone may be eligible.
    2. Subjects with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
    3. Subjects with a history of autoimmune hepatitis, systemic lupus erythematosus, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener granulomatosis, Sjögren syndrome, multiple sclerosis, or glomerulonephritis will be excluded.
    4. Subjects with a history of immune thrombocytopenic purpura, autoimmune hemolytic anaemia, Guillain-Barré syndrome, myasthenia gravis, myositis rheumatoid arthritis, vasculitis, or other autoimmune diseases will be excluded unless they have not required systemic therapy in the last 12 months.
32. Subject with history of confirmed progressive multifocal leukoencephalopathy (PML)
33. Active malignancy other than the one treated in this research. Prior history of malignancies unless the subject has been free of the disease for ≥ 2 years. However, subjects with the following history/concurrent conditions are allowed:

    1. Basal or squamous cell carcinoma of the skin
    2. Carcinoma in situ of the cervix
    3. Carcinoma in situ of the breast
    4. Incidental histologic finding of prostate cancer (T1a or T1b) using the tumor, nodes, metastasis [TNM] clinical staging system.
34. Pregnant, planning to become pregnant or lactating WOCBP.
35. Any significant medical conditions, laboratory abnormality or psychiatric illness likely to interfere with participation or understanding of study requirements (according to the investigator's decision).
36. Severe or debilitating pulmonary disease, history of interstitial lung disease, noninfectious pneumonitis, or uncontrolled lung diseases, including but not limited to pulmonary fibrosis and acute lung diseases.
37. Known or suspected history of HLH unless related to lymphoma.
38. Clinically significant history of cirrhotic liver disease, ongoing, drug-induced liver injury, alcoholic liver disease, nonalcoholic steatohepatitis, primary biliary cirrhosis, ongoing extrahepatic obstruction caused by cholelithiasis, cirrhosis of the liver, or portal hypertension.
39. INR or PT > 1.5 x ULN, or Quick percentage < 70% (if Quick percentage used in lieu of time-based units for reporting PT), in the absence of therapeutic anticoagulation.
40. aPTT >1.5 x ULN in the absence of therapeutic anticoagulation or a lupus anticoagulant.
41. Prior solid organ transplantation.
42. Person deprived of his/her liberty by a judicial or administrative decision.
43. Person hospitalized without consent.
44. Adult person under legal protection.

NB: for 42, 43, 44 if there is an individual benefit for such subjects, an Ethics Committee will have to be informed case by case.

-

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
PFS at the end of C17 (each cycle is 21 days) | end of cycle 17 (each cycle is 21 days)
  The primary efficacy endpoint is the PFS at 12 months (end of C17) from first dose of study treatment, in each cohort: Zanubrutinib/Venetoclax/Glofitamab for cohorts A and C, Venetoclax/Glofitamab for cohort B, as determined by imaging central review (Lugano 2014 criteria),

SECONDARY OUTCOMES:
Overall Response Rate (ORR) and Complete Response Rate (CRR) | End of C3 (each cycle is 21 days), end of C6 (each cycle is 21 days), end of C12 (each cycle is 21 days), end of C17 (each cycle is 21 days), end of C26 (each cycle is 21 days))
  ORR and CRR as determined by PET-CT evaluation according to Lugano 2014 (imaging central review and local assessment) and at end of C35 (24 months) determined by CT-scan only
PFS at the end of C17 as determined by investigator | end of cycle 17 (each cycle is 21 days)
  PFS at 12 months (end of C17) from first dose of study treatment as determined by investigator (Lugano 2014 criteria
Duration of response (DOR) | 72 months
  Duration of response (DOR) as determined by investigator (Lugano 2014 criteria) defined as time from first documented Complete Response or Partial Response to date of disease progression or death,
Event-free survival (EFS) | 74 months
  Event-free survival (EFS) as determined by investigator (Lugano 2014 criteria) defined as time from first dose of study treatment to earliest of: progression, next anti-lymphoma treatment, or death.
Disease Free Survival (DFS) | 74 months
  Disease Free Survival (DFS) as determined by investigator (Lugano 2014 criteria) defined as time from first dose of study treatment to earliest of: progression, or death from lymphoma.
Overall Survival (OS) | 74 months or death
  Overall survival defined as time from first dose of study treatment to death from any cause,
Time to next anti-lymphoma treatment (TTNT) | date of next anti-lymphoma treatment (74 months)
  Time to next anti-lymphoma treatment (TTNT) defined as time from first dose of study treatment to earliest date of next anti-lymphoma treatment (except corticosteroids)
Safety and tolerability: | from ICF signature until 28 days after the last treatment administration
  Incidence of grade ≥3 adverse events, adverse events of special interest (AESI).
Minimal Residual Disease (MRD) | before Cycle 1 Day1 (baseline), end of C3 (each cycle is 21 days), end of C6 (each cycle is 21 days), end of C17 (each cycle is 21 days)
  MRD response

CONTACTS AND LOCATIONS:
Overall Officials: Steven LE GOUILL, Pr, Study Chair — Institut Curie; Clementine SARKOZY, MD, Study Chair — Institut Curie; Louise ROULIN, MD, Study Chair — Hôpital Henri-Mondor - AP-HP; Gilles CROCHET, MD, Study Chair — CHU Dinant Godinne UCL Namur - YVOIR
Locations (16):
- Belgium (4):
  - Az Sint-Jan Brugge - Oostende Av, Bruges
  - Institut Jules Bordet, Brussels
  - Chu de Liege, Liège
  - Chu Ucl Namur - Site Godinne, Yvoir
- France (12):
  - Aphp - Hopital Henri Mondor, Créteil
  - Chu Dijon Bourgogne, Dijon
  - Chu de Lille - Hopital Claude Huriez, Lille
  - Institut Paoli Calmettes, Marseille
  - Chu de Montpellier, Montpellier
  - Chu de Nantes, Nantes
  - Chu Lyon-Sud, Pierre-Bénite
  - Chu de Reims - Hopital Robert Debre, Reims
  - Chu Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut Curie, Saint-Cloud
  - Institut de Cancerologie Strasbourg Europe, Strasbourg

IPD SHARING:
Plan to Share IPD: No